CLINICAL TRIAL: NCT01776606
Title: Efficacy and Safety Study of Botulinum Toxin Type A for Moderate to Severe Crow's Feet Lines
Acronym: RADIANT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RT001-CL019
Record Dates: First submitted 2013-01-18; First posted 2013-01-28 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Skin Aging
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dose A (Active Comparator): Dose A: Botulinum toxin type A
  Interventions: Drug: Botulinum Toxin Type A
- Dose B (Placebo Comparator): Dose B: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Botulinum Toxin Type A, Dose A; dose applied to the lateral canthal lines
  Arms: Dose A
Drug: Placebo — Placebo, Dose B; dose applied to the lateral canthal lines
  Arms: Dose B

SUMMARY:
This study will evaluate the efficacy and safety of botulinum toxin type A compared to placebo control for the treatment of moderate to severe crow's feet lines.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe crow's feet lines
* Female or male, 18 to 65 years of age and in good general health
* Women of childbearing potential (WOCBP) must agree to use an effective method of birth control during the course of the study

Exclusion Criteria:

* Any neurological condition that may place the subject at increased risk with exposure to botulinum toxin type A
* Muscle weakness or paralysis, particularly in the area receiving study treatment
* Active skin disease or irritation at the treatment area
* Deep dermal scarring, or inability to smooth out the crow's feet lines to be treated by manually spreading the skin apart
* Treatment with botulinum toxin type A for crow's feet lines in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Composite endpoint based upon the investigator global assessment and patient assessment of severity of lateral canthal lines | Week 4

SECONDARY OUTCOMES:
Proportion of subjects with 2 point or greater improvement from baseline using the Investigator Global Assessment | Week 4
Proportion of subjects with 1 point or greater improvement from baseline using the Investigator Global Assessment | Week 4
Proportion of subjects with a 2 point or greater improvement from baseline using the Patient Severity Assessment | Week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Research Institute, Coral Gables, Florida, United States